CLINICAL TRIAL: NCT05188807
Title: The Correlation of the Cervical Symptoms With Endotracheal Intubation Quality and Preoperative Airway Assessment With Ultrasonography and Magnetic Resonants Imaging, in Patients Operated for Cervical Symptoms
Brief Title: The Correlation of the Cervical Symptoms With Intubation Quality and Airway Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Gülencan Yumuşak Ergin, Principal Investigator, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GErgin
Record Dates: First submitted 2021-12-04; First posted 2022-01-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cervical Pain; Cervical Disease
Keywords: videolaryngoscopy; quality of intubation; cervical pathology; difficult airway
MeSH Terms: conditions — Neck Pain; Uterine Cervical Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The patient with cervical pathology (Experimental): we will perform airway ultrasonography before the patients intubations and we will intubate the patients before cervical surgery
  Interventions: Diagnostic Test: Airway ultrasonography

INTERVENTIONS:
Diagnostic Test: Airway ultrasonography — we will measure hyomental distance, skin-epiglottis distance, skin-hyoid distance, epiglottis-vocalcords distance

SUMMARY:
Cervical spine disorders can cause neck pain with or without neurological dysfunction. The most common cause of acute and chronic neck pain is cervical degenerative changes. Surgical decision of cervical pathology is made by anamnesis, neurological examination and imaging methods. Airway management can be difficult for patients presenting for cervical spine surgery. In addition, these patients may have severe cervical spine instability or spinal cord level myelopathy and may develop serious neurological complications associated with the intubation technique. Videolaringoscopes, which have become widely used with the developing technology, provide a better view than direct laryngoscopy in terms of cervical immobilization during intubation. Therefore, videolaryngoscope is preferred for cervical pathologies. Nowadays, the use of videolaryngoscope is recommended in patients with airway difficulty. Neutral position is important for intubation of patients with cervical pathology and it is highly recommended in the literature to evaluate these patients as difficult airways. All cervical patients are intubated with videolaryngoscope in investigator's clinic. The aim of this study was to evaluate how long the duration of cervical pathology affects airway anatomy and how it affects airway management during anesthesia. On the other hand, airway-related measurements will be performed by MRI and ultrasonography (USG), which is routinely evaluated in the diagnosis process, and it will be aimed to evaluate these measurements in terms of their effects on intubation quality. At the end of the study, all evaluations were analyzed and it was aimed to compare the effects of other evaluated parameters (such as USG and MRI measurements) on intubation difficulty level, with cervical pathology duration being primary.

ELIGIBILITY:
Inclusion Criteria:

- Elective cervical surgery

Exclusion Criteria:

* Patients undergoing emergency surgery
* Cervical tumor patients
* Patients with cognitive dysfunction
* Patients with previous cervical surgery
* Pediatric patients
* Cervical trauma patients
* The presence of cervical spondylitis, spondylodiscitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
intubation time in seconds | 10 minutes
  for assessing the degree of difficulty in intubation

SECONDARY OUTCOMES:
distance of measurements of airway | 10 minutes
  ultrasonographic measurements such as skin epiglottis distance, skin hyoid distance, epiglottis to vocal cords distance, hyomental distance

CONTACTS AND LOCATIONS:
Overall Officials: Gulencan Yumusak Ergin, Principal Investigator — Ankara University
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No